CLINICAL TRIAL: NCT01115426
Title: Long-term Treatment by Inhibitors of Angiotensin II at Low Doses in Non-nephrotic Proteinuric Patients With Pauciimmune and IgA Mesangioproliferative Glomerulonephritis
Brief Title: Inhibitors of Angiotensin II in Proteinuric Mesangioproliferative Glomerulonephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Pierangela Presta, "Magna Graecia" University of Catanzaro, Nephrology Unit
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGAMsPGNPMsPGN
Record Dates: First submitted 2010-04-28; First posted 2010-05-04 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 1997-01

CONDITIONS: IGA Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Ramipril; Losartan; Renin-Angiotensin System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-angiotensin II drugs (Other): Never treated patients with non-nephrotic proteinuria (1-3 g/day), microhematuria, no-evidence of renal failure or other relevant diseases and with diagnosis of I-II stage IgA- or pauciimmune-MsPGN were considered eligible.
  Interventions: Drug: Ramipril or losartan

INTERVENTIONS:
Drug: Ramipril or losartan — Ramipril (5 mg/day) was started soon after the enrollment and continued throughout the follow-up, having Losartan (50 mg/day) as alternative.
  Other Names: renin-angiotensin system (RAS) inhibitors

SUMMARY:
This study evaluates prospectively the effects of an anti-angiotensin II regimen on renal outcome in patients with mesangioproliferative glomerulonephritis followed-up for 10 years.

DETAILED DESCRIPTION:
After signing informed consent, enrolled patients started treatment with ACEi. We decided to prescribe to all patients the same drug (ramipril) at the same dosage (5 mg/day). All patients were examined every 2 months during the first year of follow-up and every 6 months thereafter. At each visit, they underwent a complete physical examination. If the target blood pressure of <140/90 mmHg was not achieved with ramipril monotherapy, addition of other antihypertensive drug(s) was allowed. Patients complaining adverse side effects attributed to ramipril were switched to losartan (50 mg/day). The patients were also prescribed a normal protein (1 gram/kg/day) and moderately salt-restricted (6-8 grams/day) diet throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* proteinuria ≥ 1 g and < 3 g/24 hours stable during the 3 months of run-in
* microscopic hematuria (with at least 10 red blood cells per high-power field), without other signs or symptoms of systemic diseases stable during the 3 months of run-in
* no-evidence of renal failure or other relevant diseases
* biopsy diagnosis of I-II stage IgA- or pauciimmune-MsPGN

Exclusion Criteria:

* estimated Glomerular Filtration Rate (eGFR) <80 ml/min/1.73m2
* previous immunosuppressive treatment
* blood pressure (BP) >150/90 mmHg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1997-01; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
renal function and proteinuria | at the end of first year of observation
  In particular, the end points of the study were a loss >20% of basal GFR and a decrease of basal daily proteinuria < 20% at the end of first year of observation.
  GFR was calculated using both the abbreviated Modification of Diet in Renal Disease (MDRD) study equation and measured creatinine clearance. For each patient, a time-averaged (TA) proteinuria were calculated as an average of the mean of every-6month period's 24-hour proteinuria measurements.

SECONDARY OUTCOMES:
serum levels of creatinine | at the end of first years of observation

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Fuiano, Professor, Study Chair — "Magna Graecia" University of Catanzaro, Nephrology Unit
Locations (1):
- "Mater Domini" Hospital, Catanzaro, Calabria, Italy

REFERENCES:
- [Derived] Presta P, Minutolo R, Iodice C, Comi N, Casoria V, Fuiano L, Caglioti C, Conte G, Fuiano G. Renin-angiotensin system inhibitors reduce the progression of mesangioproliferative glomerulonephritis: 10 year follow-up. Eur J Intern Med. 2011 Dec;22(6):e90-4. doi: 10.1016/j.ejim.2011.08.021. Epub 2011 Sep 28. PMID 22075320